CLINICAL TRIAL: NCT06056271
Title: Clinical and Healthcare Outcomes From Real-World Use in the United States of a Companion AI During AF Ablation
Acronym: COMPANION AI
Status: Recruiting | Type: Observational
Sponsor: Volta Medical (Industry)
Collaborators: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: CLIPL-01-005
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: AF Ablation — Percutaneous, catheter-based ablation of atrial fibrillation

SUMMARY:
Observational, multi-center, clinical device registry for US patients with a primary goal to observe the clinical outcomes in patients who are mapped with Volta Medical's VX1 or AF-Xplorer systems during AF ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 21 years of age or older who is:

   * indicated for AF ablation or
   * Who has received an AF-ablation with the past 24 months where VX1 was used or
2. Patients are receiving or received a catheter ablation procedure for AF according to current guidelines
3. Patients must be able and willing to provide written informed consent to participate in the clinical trial

Exclusion Criteria:

1. Patients not indicated or were not indicated for catheter ablation according to current guidelines
2. Patients with AF secondary to an obvious reversible cause
3. Patients who are or may potentially be pregnant
4. Enrollment in an investigational study evaluating another non-VX1 investigational device, biologic, or drug

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients indicated for ablation for atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary Clinical Efficacy Outcome | 12 and 24 months
  Percentage of subjects free from clinically significant AF or atrial arrhythmia recurrences, after one or multiple ablation procedures, stratified by type of clinical workflow and ablation history.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Endeavor Health, Evanston, Illinois
  - Kansas City Cardiac Arrhythmia Research LLC, Overland Park, Kansas
  - Northwell Health, New York, New York
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No